CLINICAL TRIAL: NCT01467388
Title: Efficacy of Selective Laser Trabeculoplasty in Pseudophakic Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: SLT-Pseudophakic-201
Record Dates: First submitted 2011-11-03; First posted 2011-11-08 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2014-12

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: patients with glaucoma or ocular hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- phacic: Study patients who still have their own ocular lens
  Interventions: Procedure: selective laser trabeculoplasty (SLT)
- pseudophacic: Study patients who have an intraocular lens after cataract surgery
  Interventions: Procedure: selective laser trabeculoplasty (SLT)

INTERVENTIONS:
Procedure: selective laser trabeculoplasty (SLT) — trabeculoplasty with an SLT-Laser to reduce intraocular pressure
  Other Names: SLT-Laser, Tango Laser, Ellex Medical Pty. Ltd., 82 Gilbert Street, Adelaide, SA 5000 Australia

SUMMARY:
Retrospective analysis of efficacy of selective laser trabeculoplasty in pseudophakic patients compared to phakic patients is performed.

Inclusion criterion are patients with glaucoma or ocular hypertension who underwent treatment with selective laser trabeculoplasty due to insufficient control of intraocular pressure during their routine treatment at the University Hospital Zurich / Division of Ophthalmology.

ELIGIBILITY:
Inclusion criteria:

* Patients with glaucoma or ocular hypertension who underwent selective laser trabeculoplasty.

Exclusion criteria:

* Optic neuropathy other than glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: glaucoma patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-11; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
IOP | t0

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich; Jens Funk, Professor, MD, Principal Investigator — University Hospital Zurich, Ophtalmic Clinic
Locations (1):
- University Hospital Zurich, Ophthalmic Clinic, Zurich, Canton of Zurich, Switzerland